CLINICAL TRIAL: NCT04812652
Title: Digitally Distributed Yoga Intervention for Women Treated for Breast Cancer: Effects on Fatigue, Systemic Inflammation and Levels of Activity: A Randomized Controlled Trial
Brief Title: Digitally Distributed Yoga for Women Treated for Breast Cancer
Acronym: DigiyogaCare
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: The Swedish Breast Cancer Association (Unknown); Uppsala-Örebro Regional Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 275078
Record Dates: First submitted 2021-02-03; First posted 2021-03-23 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasm Female
Keywords: breast neoplasm; breast cancer; yoga; digital intervention; eHealth; rehabilitation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group: Digitally distributed yoga (Experimental): Type of yoga: Physical yoga sequences that through scientific evaluation have proven to be effective and relevant for the target group. There will be 3 different programs during the 12-week-intervention Dose: twice weekly for 12 weeks; one yoga class live broadcasted and digitally distributed to the patient's computer or mobile device, and one class pre-recorded video for self-training.
  Sequences: The yoga class will be 60 minutes including 10 minutes of final relaxation. Thereafter, a 5 minutes reflection will be offered.
  Home Training: Instructions for yoga home practice will be standardized. The three yoga programs will be distributed in video-links for the participants to view at a time-point that suits them during the week. The recommendation will be to yoga at home once a week in addition to the digital yoga class in real time.
  Participants are expected to use their own computer or mobile device.
  Interventions: Behavioral: Digitally distributed yoga
- Control group: Regulare care (No Intervention): Receive regular care, including written standardized information about the importance of physical activity by their contact nurse or physiotherapist, when discharged from the hospital accordingly to the routines at the clinic.

INTERVENTIONS:
Behavioral: Digitally distributed yoga — Yoga distributed through internet.
  Other Names: DigiYogaCaRe
  Arms: Intervention group: Digitally distributed yoga

SUMMARY:
Breast cancer is the most common cancer disease in women. As the prevalence of fatigue is high in this group it is motivated to find interventions that can reduce fatigue and render in an increased level of physical activity both during and after treatment. Yoga have shown effect on cancer related fatigue (CRF) and is a rehabilitation activity that is often requested by breast cancer patients. Breast cancer patients live in cites and small-towns as well as in rural areas and therefore there is a need for accessible rehabilitation activities for all patients despite place of residence.

A digitally distributed yoga class can potentially increase accessibility for those living in rural areas.

Aim

The overarching aim of this study is to investigate the effect of a 12-weeks digitally distributed yoga intervention for women treated for breastcancer, compared with a control group receiving regular care, concerning:

* patient reported outcomes, primary endpoint CRF
* systemic inflammation
* activity level

The study will evaluate if there are differences during and after the intervention and if those differences are sustained after 1, 3, 6, 12 and 24 months after the intervention.

Additional objectives are to compare the two groups concerning completing oncologic treatment, cost effectiveness, return to work and also to describe the patients experiences of participating in a digitally distributed yoga class at home.

Research questions

If and how a digitally distributed yoga can influence cancer related fatigue, stress, health related quality of life and level of physical activity compared to regular care? If and how a digitally distributed yoga can have an effect on systemic inflammation? How is the feasibility of digitally distributed yoga twice weekly at home? What is the breast cancer patients' experience of participating in digitally distributed yoga clas?

DETAILED DESCRIPTION:
Study design and Setting

This is a randomized controlled multi center study where the participant are randomized to a 12-weeks internet based yoga intervention or regular care. Usual care includes standardized information about the importance of physical activity in their personal care plan.

Three regions located in the middle of Sweden is reqruiting participants and two moore is in the process of starting reqruitment.

From January 2022 permission to reqruit through social media and direct adverticement began, after permission was granted from the ethical board.

Inclusion criteria: Adult women diagnosed with breast cancer, that have undergone breast cancer surgery within 60 days with curative intention, without any signs of metastatic disease, and before start of chemotherapy. They should be Swedish speaking and literate.

Exclusion criteria: If they received neoadjuvant treatment before surgery, have an advanced recurrent disease, unstable cardiovascular disease, brain or bone metastasis or are unable to complete the questionnaires due to reduced physical or cognitive capacity. If they have any physical condition that hinder participation in yoga or have an unstable medical condition that might be aggravated by yoga.

Randomization:

The patients are randomized after their first visit to the oncologist. In an web-based digital portal, a digital randomization are conducted. The stratified randomization will be according to surgery, Breast-Conserving Surgery (BCS) versus mastectomy (ME), chemotherapy versus no chemotherapy.

Yoga Intervention:

To minimize the ambiguities in design found in previous studies, the yoga intervention is designed according to Sherman's recommendations. The yoga postures and movements will be chosen specifically to address this group of patients.

1. Type of yoga: Physical yoga sequences that through scientific evaluation have proven to be effective and relevant for the target group, ended by relaxation and time for reflection. There are two different programs during the 12-week-intervention. Easy-access sequences that can suit all (with modifications if needed), no progression but the programs can offer a small variation of movements over the intervention period.
2. Dose: twice weekly for 12 weeks; one yoga class live broadcasted and digitally distributed to the patient's computer or mobile device, and one class pre-recorded video for self-training.
3. Components of yoga: The yoga class will follow a standardized program with yoga sequences that is designed to increase calm, improve focus, acceptance and energy level as well as reduce fatigue.
4. Sequences: The yoga class will be 60 minutes including 10 minutes of final relaxation. Thereafter, a 5 minutes reflection will be offered.
5. Modification: Modification of yoga movements will be offered by the instructors based on the personal conditions of the participants. In the pre-recorded video the instructor will give a number or alternatives when relevant.
6. Selection of instructors: The yoga instructors have previous experience of teaching yoga, ie is registered yoga teachers with 100 respectively 200-hour training. They have attend a one-day course administered by the research team consisting of lectures and seminars about cancer and cancer treatment, the aim and design of the study, theory, and instructions regarding the yoga programs including modifications and technical aspects regarding digital distribution of the intervention.
7. Home Training: Instructions for yoga home practice will be standardized. The yoga programs will be distributed in video-links for the participants to view at a time-point that suits them during the week. The recommendation will be to yoga at home once a week in addition to the digital yoga class in real time.
8. Presence over time: Attendance will be noted through login data. Adherence to activity will be calculated as the number of patients conducting 65% of the sessions, divided by the total number of patients in the group.

Technical solution:

Participants are expected to use their own computer or mobile device. The streaming is be arranged through Zoom® . Written information and help to connect is provided weekly as well as personal support when needed.

Control group:

All breast cancer patients receives written standardized information about the importance of physical activity by their contact nurse or physiotherapist, when discharged from the hospital accordingly to the routines at the clinic.

Sample size estimation:

The sample size calculation is based on the outcome fatigue. The target main effect size is determined to be an improved fatigue score of 2 on a scale from 4 to 20. That is in accordance with the clinical important difference. For two-sided test with α=0.05 and power =80% to detect a factorial effect of 2 under the null hypothesis of no effect, 64 individuals in each group are needed. In order to compensate for a potential 30% dropout, the sample size will be increased with an additional 39 persons, giving a total sample size of 67 patients. To detect interaction effects that is usually smaller than the main effect, the original sample size was increased with 25% (~42 patients). This gives a total of 209 patients divided into 2 arms; intervention and control. To cover up for any other possible dropouts a total of 240 perons will be included.

Data collection:

Data are collected at baseline (one month after surgery) and 3, 6, 24 and 48 months after breast cancer surgery. Self-reported data (questionnaires) are collected each time (5 times), activity levels (accelerometer) at the first three follow-ups and at 12 months.

Diary of physical activity is reported in conjunction with the measurements with accelerometer.

Blood samples will be collected from 40 patients reqruited through hospitals at the first three follow-ups.

Health economic evaluation:

The health economic evaluation will be performed with a societal as well as a health care perspective and consider time period from baseline to one year after the interventions had ended. Cost effectiveness will be presented in costs per quality adjusted life years (QALY), but also as a probability of cost-effectiveness compared to usual care.

Main components in the analysis are extra costs of the interventions, changes in QALY and savings of the interventions. Saving may be less time on sick leave (less production losses) and less health care consumption. Complete costs of the interventions for the health care provider and for patients will be measured. Further, QALY will be estimated using the instrument EQ-5D-5L, time on sick leave will be collected in the questionnaire to participants, and health care consumption will be retrieved from medical records.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosed with breast cancer Adult women Must have undergone breast cancer surgery with curative intention Must be Swedish speaking Must be able to read

-

Exclusion criteria:

Metastatic disease Received neoadjuvant treatment before surgery Advanced recurrent disease Unstable cardiovascular disease Brain or bone metastasis Unstable medical condition that might be aggravated by yoga.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 229 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cancer related fatigue | Baseline is 1 months after surgery and change after 3, 6, 24 and 48 months after breast cancer surgery
  The Multidimensional Fatigue inventory (MFI) is a 20-item self-reported questionnaire including 5 subscales: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation is a state of physical, emotional, cognitive tiredness or exhaustion related to cancer. The score can be between 20 and 100. Higher score indicate higher fatigue.

SECONDARY OUTCOMES:
Change in Stress | Baseline is 1 months after surgery and change after 3, 6, 24 and 48 months after breast cancer surgery
  Instrument:The Perceived Stress Scale (PSS) measures general stress and coping capabilities. The instrument is validated on a Swedish population and has 14 questions. There are 4 alternative to each item. A higher score indicates higher stress. Each item minimum 0 and maximum 4
Change in Health related Quality of Life (HRQoL) | Baseline is 1 months after surgery and change after 3, 6, 24 and 48 months after breast cancer surgery
  Instrument: European Organization for Research and Treatment of Cancer EORTC-QLQ30 . Measures generic HRQoL and comprises 30 items grouped into six multi-item scales: Global health status, Physical functioning, Role functioning, Emotional functioning, Cognitive functioning and Social functioning. Inclusive symptom scales,; nausea, pain, dyspnea , insomnia, loss of apatite, constipation and diarrhea.
  Breast-23 is the breast cancer specific module for EORTC in breast cancer patients with additional 23 items.
  A higher score in Global health status and functioning scales indicates higher HRQL while high values in symptom scores indicates high symptom burden. Minimum is 0 and maximum is 100.
Change in Quality of life | Baseline is 1 months after surgery and change after 3, 6, 24 and 48 months after breast cancer surgery
  Instrument: The EuroQol 5-dimensions is a generic standardized instrument to measure HRQoL in health economic analysis. The instrument includes five dimensions; mobility, self-care, usual activities, pain/discomfort and anxiety/depression and includes five response levels; no problems, slight problems, moderate problems, severe problems, unable to/extreme problems . Minimum 0 and maximum 4. Low values indicates higher quality of Life.

OTHER OUTCOMES:
Changes in physical activity | Baseline is 1moths after surgery and changes at 3, 6 and 12 months after surgery
  Physical activity: will be measured to be able to see changes in activity level that may be an effect of reduced fatigue and increased energy level. Measurement is carried out with an accelerometer (advanced pedometer ) for 7 days on 4 Occasion. Data on physical activity will be combined with body weight to calculate energy expenditure complemented with a diary for the same time period that describes the type of activity
Changes in IL-1 | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Pro-inflammatory marker; blood sample
Diagnose related measurement: Side effects | After one and two year.
  Side effects from cancer treatment will be collected according to National Cancer Institute Common Toxicity Criteria.
Rate of Sick Days | One and two years after the intervention
  From the Statistical and result database (STORE), managed by the Swedish Social Security Agency, data of sick days will be collected.
Changes in IL-1β, | Baseline is 1 months after surgery and changes are measured at 3 and 6 months
  Pro-inflammatory marker
Changes in IL-8 | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Pro-inflammatory marker , blood sample
Changes in IL-12 | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Pro-inflammatory marker , blood sample
Changes in Serum Hs | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Inflammatory marker, blood sample
Changes in C reactive protein | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Inflammatory marker,blood sample
Changes in Tumor necrosis factor -α | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Inflammatory markers, blood sample
Changes in sTNFRII, | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Inflammatory marker, blood sample
Changes in Fibrinogen | Baseline is 1 months after surgery and changes are measured at 3 and 6 months after surgery
  Inflammatory marker, blood sample
Changes in IGF-1 | Baseline is 1 months after surgery and changes are measured at 3 and 6 months
  Metabolic marker, blood sample
Changes in Insulin-like growth factor II (IGF-II), | Baseline is 1 months after surgery and changes are measured at 3 and 6 months
  Metabolic marker, blood sample
Changes in Leptin | Baseline is 1 months after surgery and changes are measured at 3 and 6 months
  Metabolic marker, blood sample
Changes in Adiponectin | Baseline is 1 months after surgery and changes are measured at 3 and 6 months
  Metabolic marker,blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Emma Ohlsson-Nevo, PH.D, Study Chair — University Healthcare Research Center, Region Örebro County, Sweden
Locations (3):
- Sweden (3):
  - Gävle sjukhus, Gävle
  - University Health Care Center, Örebro
  - Västmanlands Hospital, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohlsson Nevo E, Arvidsson-Lindvall M, Hellerstedt Borjeson S, Hagberg L, Hultgren Hornqvist E, Valachis A, Wickberg A, Duberg A. Digitally distributed Yoga Intervention in Breast Cancer Rehabilitation (DigiYoga CaRe): protocol for a randomised controlled trial. BMJ Open. 2022 Nov 1;12(11):e065939. doi: 10.1136/bmjopen-2022-065939. PMID 36319059
- [Derived] Nilsson MB, Arvidsson Lindvall M, Fesse PWT, Hellerstedt-Borjesson S, Ohlsson-Nevo E, Duberg A. Experiences of Home-Based Participation in a Digitally Distributed Yoga Intervention in Breast Cancer Rehabilitation: Qualitative Content Analysis. J Med Internet Res. 2025 Nov 20;27:e75975. doi: 10.2196/75975. PMID 41264913
- [Derived] Messer S, Oeser A, Wagner C, Wender A, Cryns N, Scherer RW, Mishra SI, Monsef I, Holtkamp U, Andreas M, Brockelmann PJ, Ernst M, Skoetz N. Yoga for fatigue in people with cancer. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015520. doi: 10.1002/14651858.CD015520. PMID 40421669